CLINICAL TRIAL: NCT05363358
Title: Evaluating the Safety of GAMMAGARD LIQUID for the Treatment of Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Brief Title: A Safety Study of GAMMAGARD LIQUID (GGL) in Participants With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry); RTI Health Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: TAK-771-4002; EUPAS46101 (Other: EUPAS)
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ig-naive (New-to-class) Cohort: Participants who initiate GGL or one of the comparator IVIG products who have no record of previous use of any Ig product (Ig naive) for at least 6 months before study initiation will be include in this cohort.
- Ig-experienced (New-to-drug) Cohort: Participants who initiate either GGL or a comparator IVIG product with no record of previous use of that specific IVIG product but with previous use of any other Ig product (Ig experienced) in all available study data will be included in this cohort.

SUMMARY:
The main aim of this study is to evaluate the rates of adverse events of special interest (AESIs) (thrombotic events, acute kidney injury [AKI], and hemolytic events) among participants with CIDP initiating GGL compared with rates among participants with CIDP initiating comparator intravenous immunoglobulin (IVIG) products.

No study medicines will be provided to participants in this study.

ELIGIBILITY:
Inclusion Criteria:

* Have a minimum of 6 months of continuous enrollment in the study database with medical and pharmacy coverage before the index date. Gaps in continuous enrollment less than or equal to (<=) 31 days are permitted.
* Fulfill the Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) diagnosis algorithm on or before the index date using all available baseline data for each participant.
* Additionally, to be eligible for the Ig-naive (new-to-class) cohort, participants will be required to meet the following inclusion criterion:
* Be free of any previous recorded use of any Ig product at any point before IVIG initiation.
* To be eligible for the Ig-experienced (new-to-drug) cohort, participants will be required to meet the following inclusion criterion:
* Have any previous recorded use of an Ig product at any point before the index date.

Exclusion Criteria:

* Having claims for greater than or equal to (>=) 2 different IVIG products on the index date.
* Recorded diagnosis of any of the following conditions where Ig products are used for treatment on or before the index date

  1. Primary immunodeficiency disease (PID).
  2. Evidence of secondary immunodeficiency (SID), including hematological malignancy (e.g., diagnosis of multiple myeloma or chronic lymphocytic leukemia) or treatment with rituximab.
  3. Idiopathic thrombocytopenic purpura (ITP).
  4. Dermatomyositis or polymyositis.
  5. Systemic sclerosis/scleroderma.
  6. Myasthenia gravis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CIDP on treatment with GGL and other IVIG products will be observed in this retrospective study.
Sampling Method: Non-Probability Sample
Enrollment: 6086 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Thrombotic Events (TEs) | Throughout observational period, from 01 January 2008 to 31 December 2019 (Up to 12 years)
  Thrombotic events will be reported as adverse events of special interest (AESI) and will include: acute ischemic stroke, acute myocardial infarction (AMI), and acute venous thromboembolism (VTE) events including (deep vein thrombosis (DVT), cerebral venous thrombosis (CVT), pulmonary embolism (PE).
Number of Participants With Acute kidney injury (AKI) | Throughout observational period, from 01 January 2008 to 31 December 2019 (Up to 12 years)
  AKI will be reported as AESI and will include acute renal failure.
Number of Participants With Hemolytic Events (HEs) | Throughout observational period, from 01 January 2008 to 31 December 2019 (Up to 12 years)
  HEs will be reported as AESI and will include nonautoimmune hemolytic anemia, acquired hemolytic anemia, ABO incompatibility reaction, or hemolytic transfusion reaction.

SECONDARY OUTCOMES:
Number of Participants With Anaphylaxis | Throughout observational period, from 01 January 2008 to 31 December 2019 (Up to 12 years)
  Anaphylaxis will be reported as adverse event (AE) and will include anaphylactic reaction or anaphylactic shock.
Number of Participants With Transfusion-related Acute Lung Injury (TRALI) | Throughout observational period, from 01 January 2008 to 31 December 2019 (Up to 12 years)
  Number of participants with TRALI will be reported.
Number of Participants With Transfusion-associated Circulatory Overload (TACO) | Throughout observational period, from 01 January 2008 to 31 December 2019 (Up to 12 years)
  Number of participants with TACO will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- RTI Health Solutions, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/efe528d2b61341d9?idFilter=%5B%22TAK-771-4002%22%5D